CLINICAL TRIAL: NCT03817125
Title: A Multicenter Phase 1b Randomized, Placebo-controlled, Blinded Study to Evaluate the Safety, Tolerability and Efficacy of Microbiome Study Intervention Administration in Combination With Anti-PD-1 Therapy in Adult Patients With Unresectable or Metastatic Melanoma
Brief Title: Melanoma Checkpoint and Gut Microbiome Alteration With Microbiome Intervention
Acronym: MCGRAW
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parker Institute for Cancer Immunotherapy (Other)
Collaborators: Seres Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PICI0014
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma; anti-PD1; Nivolumab; Microbiome; SER-401
MeSH Terms: conditions — Melanoma | interventions — Anti-Bacterial Agents; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomly assigned in a 2:1 ratio to oral microbiome study intervention or matching placebo. Nivolumab will be administered open-label as standard of care to all groups. Investigators, site personnel, and participants will remain blinded to the assignment of microbiome study intervention throughout the course of the study. Select Sponsor personnel, including but not limited to the Medical Monitor, Clinical Scientists, Biostatistician, and Patient Safety, will be unblinded to treatment assignment for ongoing safety monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SER-401 Matching Placebo/ Nivolumab (Placebo Comparator): Participants will undergo a 4-day lead-in pretreatment with antibiotic placebo, then matching placebo for SER-401 and nivolumab (480 mg) treatment.
  Interventions: Drug: Placebo for antibiotic; Drug: Nivolumab; Drug: Matching Placebo for SER-401
- SER-401/ Nivolumab (Experimental): Participants will undergo a 4-day lead-in pretreatment with antibiotic (vancomycin) to prime the gut microbiome for engraftment of the oral microbiome study intervention, then SER-401 and nivolumab treatment.
  Interventions: Drug: Vancomycin pretreatment; Drug: Nivolumab; Drug: SER-401

INTERVENTIONS:
Drug: Placebo for antibiotic — Placebo for antibiotic will be administered orally four times a day for 4 days, followed by a 2-3 day washout.
  Arms: SER-401 Matching Placebo/ Nivolumab
Drug: Vancomycin pretreatment — Vancomycin (125mg) will be administered orally four times a day, followed by a 2-3 day washout.
  Arms: SER-401/ Nivolumab
Drug: Nivolumab — Nivolumab (480 mg) will be administered intravenously (IV) according to institutional guidelines every 4 weeks for up to 12 cycles. A cycle is defined as 4 calendar weeks.
  Other Names: Opdivo
Drug: Matching Placebo for SER-401 — Administered once a day for 7 days during the lead-in phase, followed by once a day for 8 weeks during the microbiome/anti-PD-1 treatment phase.
  Arms: SER-401 Matching Placebo/ Nivolumab
Drug: SER-401 — Administered once a day for 7 days during the lead-in phase, followed by once a day for 8 weeks during the microbiome/anti-PD-1 treatment phase.
  Arms: SER-401/ Nivolumab

SUMMARY:
This study is designed to evaluate the safety and tolerability of treatment with oral microbiome study intervention (SER-401) or matching placebo in combination with anti-programmed cell death 1 (anti-PD-1) therapy (nivolumab) in participants with unresectable or metastatic melanoma. The study also intends to assess clinical outcomes, the impact of microbiome study intervention administration on the microbiome profile, and its association with clinical and immunological outcomes.

DETAILED DESCRIPTION:
This is a Phase 1b, multicenter, randomized, placebo-controlled, blinded study in adult participants with anti-PD-1 therapy naïve, unresectable or metastatic melanoma to evaluate the safety and tolerability of SER-401, or matching placebo in combination with anti-PD-1 therapy (nivolumab). Prior to initiating microbiome study intervention and nivolumab, participants will undergo an antibiotic or antibiotic placebo treatment lead-in to prime the gut microbiome for engraftment of the oral microbiome study intervention. Study intervention groups will be assessed for safety, changes in the microbiome, changes in the percentage of tumoral CD8 T cells, and antitumor activity. Participants must have measurable disease that can be biopsied and consent to baseline and on-treatment biopsies, as well as stool and blood biomarker collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be willing to provide a baseline stool sample.
2. Histologically-confirmed Stage IV cutaneous melanoma or Stage III cutaneous, acral or mucosal melanoma that is judged inoperable. Participants with a history of uveal melanoma are not eligible.
3. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1; ie, defined as at least 1 lesion that can be accurately measured in at least 1 dimension [longest diameter to be recorded] with a minimum size of ≥ 10 mm by computerized tomography [CT] scan or caliper measurement on clinical exam or ≥ 20 mm by chest X-ray).

   1. Malignant lymph nodes must be ≥ 15 mm in short axis when assessed by CT scan to be considered pathologically enlarged and measurable.
   2. Participants must have at least one measurable lesion by RECIST and a separate lesion amenable to biopsy that has not been previously irradiated.

   i. Participants must be willing to undergo a newly-obtained core needle or incisional biopsy at baseline (prior to antibiotic or antibiotic placebo administration). Fine needle aspiration is not acceptable.
4. Participants must be willing to undergo tumor biopsy on treatment.
5. Prior adjuvant or neoadjuvant melanoma therapy is permitted if completed at least 6 weeks prior to randomization and all related AEs have either returned to baseline or stabilized.

   1. Prior anti-CTLA-4 therapy in the adjuvant setting is allowed if completed at least 12 weeks prior to the first dose of anti-PD-1.

Exclusion Criteria:

1. Participants who require hemodialysis.
2. Participants with a history of another cancer in the last 5 years, except for: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; c) localized prostate cancer not requiring systemic therapy; and c) other primary tumors with no known active disease present that, in the opinion of the Investigator and the Sponsor, will not affect participant outcome in the setting of the current diagnosis.
3. Any known, untreated brain metastases. Participants with brain metastases are eligible if these have been treated, and provided:

   1. Brain metastases must be stable (image-documented) 4 weeks after completion of treatment for brain metastases and require treatment with less than 10 mg/day prednisone equivalent for at least 2 weeks prior to study intervention administration.
   2. Neurological symptoms should be absent or returned to baseline.
4. Prior checkpoint inhibitor therapy with anti-PD-1 or anti-PD-L1 in the adjuvant setting.

   a. Exception: Participants with stage 3 or 4 cutaneous melanoma status post-resection who have received up to one year of adjuvant anti-PD-1 therapy who have recurred > 6 months after their last dose of anti-PD-1 therapy are eligible.
5. Other prior systemic treatment (ie, anticancer chemotherapy, immunotherapy, or investigational agents) for unresectable or metastatic melanoma EXCEPT:

   1. Prior BRAF-targeted therapy (ie, BRAF or BRAF-MEK) in the metastatic setting is allowed if completed at least 4 weeks prior to the first dose of anti-PD-1.
   2. Prior anti-CTLA 4 therapy in the adjuvant setting are allowed if completed at least 12 weeks prior to the first dose of anti-PD-1.
6. History of active inflammatory bowel disease (eg, active Crohn's disease or ulcerative colitis) with diarrhea OR major gastrointestinal surgery (not including appendectomy or cholecystectomy) within 3 months of enrollment (ie, signed informed consent for the study), OR any history of total colectomy or bariatric surgery (bariatric surgery which does not disrupt the gastrointestinal lumen, ie, restrictive procedures such as banding, are permitted).
7. Any diagnosis of autoimmune disease. Participants with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, adrenal insufficiency on replacement dose steroids, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

   a. Participants with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
8. Has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study intervention administration or has a contrast allergy requiring premedication with corticosteroids. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
9. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (ie, bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan.

   a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
10. Has a transplanted organ or has undergone allogeneic bone marrow transplant.
11. Has received a live vaccine within 30 days prior to first dose. Participants must not receive live, attended influenza vaccine (eg, FluMist) within 30 days prior to Cycle 1, Day 1 or at any time during the study and 100 days after last dose of nivolumab.
12. Has used antibiotics within 30 days prior to randomization or has planned or required need for antibiotic prophylaxis for more than 24 consecutive hours during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parker Institute for Cancer Immunotherapy, Study Director — Parker Institute for Cancer Immunotherapy
Locations (7):
- United States (7):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alang N, Kelly CR. Weight gain after fecal microbiota transplantation. Open Forum Infect Dis. 2015 Feb 4;2(1):ofv004. doi: 10.1093/ofid/ofv004. eCollection 2015 Jan. PMID 26034755
- [Background] Balch CM, Gershenwald JE, Soong SJ, Thompson JF, Ding S, Byrd DR, Cascinelli N, Cochran AJ, Coit DG, Eggermont AM, Johnson T, Kirkwood JM, Leong SP, McMasters KM, Mihm MC Jr, Morton DL, Ross MI, Sondak VK. Multivariate analysis of prognostic factors among 2,313 patients with stage III melanoma: comparison of nodal micrometastases versus macrometastases. J Clin Oncol. 2010 May 10;28(14):2452-9. doi: 10.1200/JCO.2009.27.1627. Epub 2010 Apr 5. PMID 20368546
- [Background] Choi HH, Cho YS. Fecal Microbiota Transplantation: Current Applications, Effectiveness, and Future Perspectives. Clin Endosc. 2016 May;49(3):257-65. doi: 10.5946/ce.2015.117. Epub 2016 Mar 9. PMID 26956193
- [Background] Dubberke ER, Lee CH, Orenstein R, Khanna S, Hecht G, Gerding DN. Results From a Randomized, Placebo-Controlled Clinical Trial of a RBX2660-A Microbiota-Based Drug for the Prevention of Recurrent Clostridium difficile Infection. Clin Infect Dis. 2018 Sep 28;67(8):1198-1204. doi: 10.1093/cid/ciy259. PMID 29617739
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Ekwueme DU, Guy GP Jr, Li C, Rim SH, Parelkar P, Chen SC. The health burden and economic costs of cutaneous melanoma mortality by race/ethnicity-United States, 2000 to 2006. J Am Acad Dermatol. 2011 Nov;65(5 Suppl 1):S133-43. doi: 10.1016/j.jaad.2011.04.036. PMID 22018062
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Background] Hamilton MJ, Weingarden AR, Unno T, Khoruts A, Sadowsky MJ. High-throughput DNA sequence analysis reveals stable engraftment of gut microbiota following transplantation of previously frozen fecal bacteria. Gut Microbes. 2013 Mar-Apr;4(2):125-35. doi: 10.4161/gmic.23571. Epub 2013 Jan 18. PMID 23333862
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Khanna S, Button JE, Lombardo MJ, Vulic M, Henn MR, Cook DN, Pomerantz RJ, Hohmann EL. Reply to Lagier et al. J Infect Dis. 2017 Jan 1;215(1):162-164. doi: 10.1093/infdis/jiw490. Epub 2016 Oct 20. No abstract available. PMID 28077592
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Lee CH, Steiner T, Petrof EO, Smieja M, Roscoe D, Nematallah A, Weese JS, Collins S, Moayyedi P, Crowther M, Ropeleski MJ, Jayaratne P, Higgins D, Li Y, Rau NV, Kim PT. Frozen vs Fresh Fecal Microbiota Transplantation and Clinical Resolution of Diarrhea in Patients With Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2016 Jan 12;315(2):142-9. doi: 10.1001/jama.2015.18098. PMID 26757463
- [Background] Lynch SV, Pedersen O. The Human Intestinal Microbiome in Health and Disease. N Engl J Med. 2016 Dec 15;375(24):2369-2379. doi: 10.1056/NEJMra1600266. No abstract available. PMID 27974040
- [Background] Matson V, Fessler J, Bao R, Chongsuwat T, Zha Y, Alegre ML, Luke JJ, Gajewski TF. The commensal microbiome is associated with anti-PD-1 efficacy in metastatic melanoma patients. Science. 2018 Jan 5;359(6371):104-108. doi: 10.1126/science.aao3290. PMID 29302014
- [Background] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):987-994. doi: 10.1093/cid/ciy149. PMID 29562266
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Paramsothy S, Kamm MA, Kaakoush NO, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Paramsothy R, Xuan W, Lin E, Mitchell HM, Borody TJ. Multidonor intensive faecal microbiota transplantation for active ulcerative colitis: a randomised placebo-controlled trial. Lancet. 2017 Mar 25;389(10075):1218-1228. doi: 10.1016/S0140-6736(17)30182-4. Epub 2017 Feb 15. PMID 28214091
- [Background] Pigneur B, Sokol H. Fecal microbiota transplantation in inflammatory bowel disease: the quest for the holy grail. Mucosal Immunol. 2016 Nov;9(6):1360-1365. doi: 10.1038/mi.2016.67. Epub 2016 Jul 27. PMID 27461176
- [Background] Qazi T, Amaratunga T, Barnes EL, Fischer M, Kassam Z, Allegretti JR. The risk of inflammatory bowel disease flares after fecal microbiota transplantation: Systematic review and meta-analysis. Gut Microbes. 2017 Nov 2;8(6):574-588. doi: 10.1080/19490976.2017.1353848. Epub 2017 Sep 12. PMID 28723262
- [Background] Ribas A, Hamid O, Daud A, Hodi FS, Wolchok JD, Kefford R, Joshua AM, Patnaik A, Hwu WJ, Weber JS, Gangadhar TC, Hersey P, Dronca R, Joseph RW, Zarour H, Chmielowski B, Lawrence DP, Algazi A, Rizvi NA, Hoffner B, Mateus C, Gergich K, Lindia JA, Giannotti M, Li XN, Ebbinghaus S, Kang SP, Robert C. Association of Pembrolizumab With Tumor Response and Survival Among Patients With Advanced Melanoma. JAMA. 2016 Apr 19;315(15):1600-9. doi: 10.1001/jama.2016.4059. PMID 27092830
- [Background] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- [Background] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Arance A, Schmidt H, Schadendorf D, Gogas H, Lundgren-Eriksson L, Horak C, Sharkey B, Waxman IM, Atkinson V, Ascierto PA. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015 Jan 22;372(4):320-30. doi: 10.1056/NEJMoa1412082. Epub 2014 Nov 16. PMID 25399552
- [Background] Routy B, Le Chatelier E, Derosa L, Duong CPM, Alou MT, Daillere R, Fluckiger A, Messaoudene M, Rauber C, Roberti MP, Fidelle M, Flament C, Poirier-Colame V, Opolon P, Klein C, Iribarren K, Mondragon L, Jacquelot N, Qu B, Ferrere G, Clemenson C, Mezquita L, Masip JR, Naltet C, Brosseau S, Kaderbhai C, Richard C, Rizvi H, Levenez F, Galleron N, Quinquis B, Pons N, Ryffel B, Minard-Colin V, Gonin P, Soria JC, Deutsch E, Loriot Y, Ghiringhelli F, Zalcman G, Goldwasser F, Escudier B, Hellmann MD, Eggermont A, Raoult D, Albiges L, Kroemer G, Zitvogel L. Gut microbiome influences efficacy of PD-1-based immunotherapy against epithelial tumors. Science. 2018 Jan 5;359(6371):91-97. doi: 10.1126/science.aan3706. Epub 2017 Nov 2. PMID 29097494
- [Background] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Sivan A, Corrales L, Hubert N, Williams JB, Aquino-Michaels K, Earley ZM, Benyamin FW, Lei YM, Jabri B, Alegre ML, Chang EB, Gajewski TF. Commensal Bifidobacterium promotes antitumor immunity and facilitates anti-PD-L1 efficacy. Science. 2015 Nov 27;350(6264):1084-9. doi: 10.1126/science.aac4255. Epub 2015 Nov 5. PMID 26541606
- [Background] Tripp MK, Watson M, Balk SJ, Swetter SM, Gershenwald JE. State of the science on prevention and screening to reduce melanoma incidence and mortality: The time is now. CA Cancer J Clin. 2016 Nov 12;66(6):460-480. doi: 10.3322/caac.21352. Epub 2016 May 27. PMID 27232110
- [Background] Vermeire S, Joossens M, Verbeke K, Wang J, Machiels K, Sabino J, Ferrante M, Van Assche G, Rutgeerts P, Raes J. Donor Species Richness Determines Faecal Microbiota Transplantation Success in Inflammatory Bowel Disease. J Crohns Colitis. 2016 Apr;10(4):387-94. doi: 10.1093/ecco-jcc/jjv203. Epub 2015 Oct 29. PMID 26519463
- [Background] Wang S, Xu M, Wang W, Cao X, Piao M, Khan S, Yan F, Cao H, Wang B. Systematic Review: Adverse Events of Fecal Microbiota Transplantation. PLoS One. 2016 Aug 16;11(8):e0161174. doi: 10.1371/journal.pone.0161174. eCollection 2016. PMID 27529553
- [Background] Weingarden A, Gonzalez A, Vazquez-Baeza Y, Weiss S, Humphry G, Berg-Lyons D, Knights D, Unno T, Bobr A, Kang J, Khoruts A, Knight R, Sadowsky MJ. Dynamic changes in short- and long-term bacterial composition following fecal microbiota transplantation for recurrent Clostridium difficile infection. Microbiome. 2015 Mar 30;3:10. doi: 10.1186/s40168-015-0070-0. eCollection 2015. PMID 25825673
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Youngster I, Mahabamunuge J, Systrom HK, Sauk J, Khalili H, Levin J, Kaplan JL, Hohmann EL. Oral, frozen fecal microbiota transplant (FMT) capsules for recurrent Clostridium difficile infection. BMC Med. 2016 Sep 9;14(1):134. doi: 10.1186/s12916-016-0680-9. PMID 27609178
- See also: NCT02437487: SER-109 Versus Placebo to Prevent Recurrent Clostridium Difficile Infection (RCDI) — https://clinicaltrials.gov/ct2/show/NCT02437487
- See also: NCT02530385: Fecal Microbiota Transplant for Obesity and Metabolism — https://clinicaltrials.gov/ct2/show/NCT02530385
- See also: NCT02618187: A Study to Evaluate the Safety, Tolerability and Microbiome Dynamics of SER- 287 in Subjects With Mild-to-Moderate Ulcerative Colitis Patients — https://clinicaltrials.gov/ct2/show/NCT02618187
- See also: NCT03341143: Fecal Microbiota Transplant (FMT) in Melanoma Patients — https://clinicaltrials.gov/ct2/show/NCT03341143
- See also: NCT03353402: Fecal Microbiota Transplantation (FMT) in Metastatic Melanoma Patients Who Failed Immunotherapy — https://clinicaltrials.gov/ct2/show/NCT03353402
- See also: NCT03637803: MRx0518 and Pembrolizumab Combination Study — https://clinicaltrials.gov/ct2/show/NCT03637803
- See also: Opdivo (nivolumab) US Prescribing Information (USPI), Aug-2018 — http://www.opdivohcp.com/?cid=sem_230964&ovl=isi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Started | 6 | 8
Completed | 4 | 2
Not Completed | 2 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lack of Efficacy | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (22.31) | 66.3 (11.73) | 61.6 (17.21)
Age, Customized [Median (Full Range); unit: years] | 60.5 [26 to 81] | 64 [46 to 84] | 64 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Ruminococcaceae abundance-based metric at Screening [Count of Participants; unit: Participants] — Stool samples were required at screening to assess fecal microbiome composition of the Ruminococcaceae abundance-based metric (high, low).The test for Ruminococcaceae is a laboratory developed test. It is not an FDA-approved device, and its use is investigational. Quantitative polymerase chain reaction (qPCR) on DNA extracted from stool was performed and the Ruminococcaceae abundance-based metric was determined.
  Participants
    Low | 4 | 5 | 9
    High | 2 | 3 | 5
ECOG Performance Score at Screening [Count of Participants; unit: Participants] — The ECOG (Eastern Cooperative Oncology Group) performance status is a widely-used scale to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine the appropriate treatment and prognosis.
  Here is a brief description of the ECOG performance status:
  * 0: Fully active, able to carry on all pre-disease performance without restriction.
  * 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework or office work.
  Participants
    0 | 6 | 7 | 13
    1 | 0 | 1 | 1
Cancer Stage at Initial Diagnosis [Count of Participants; unit: Participants] — The stage of cancer at initial diagnosis provides vital information about the extent of cancer in the body and is pivotal for prognosis and treatment decisions. Cancer stages typically range from stage 0 (in situ, localized growth) to stage IV (advanced cancer with distant metastasis).
  Participants
    IIA | 0 | 2 | 2
    IIC | 2 | 2 | 4
    IIIA | 1 | 0 | 1
    IIIB | 1 | 1 | 2
    IIIC | 0 | 2 | 2
    IV | 1 | 1 | 2
    Unknown | 1 | 0 | 1
Cancer Stage at Enrollment [Count of Participants; unit: Participants] — The stage of cancer at study enrollment provides vital information about the extent of cancer in the body and is pivotal for prognosis and treatment decisions. Cancer stages typically range from stage 0 (in situ, localized growth) to stage IV (advanced cancer with distant metastasis).
  Patients for this study needed to have histologically-confirmed Stage IV cutaneous melanoma or Stage III cutaneous, acral or mucosal melanoma that is judged inoperable by the treating physician.
  Participants
    IIIA | 1 | 0 | 1
    IIIB | 1 | 0 | 1
    IIIC | 1 | 2 | 3
    IV | 3 | 6 | 9
Melanoma Subtype [Count of Participants; unit: Participants]
  Acral | 1 | 0 | 1
  Cutaneous | 3 | 7 | 10
  Mucosal | 1 | 0 | 1
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Events (AEs)
Description: Investigators recorded AEs during each participant interaction. Symptoms were evaluated by the Investigator using the CTCAE version 5.0. This system grades AEs on a 1 to 5 scale: Grades 1 and 2 indicate mild to moderate events; Grade 3 denotes severe events; Grades 4 and 5 signify life-threatening or fatal outcomes.
  A treatment-emergent adverse event (TEAE) is defined as any event that either occurs after the initiation of study intervention, having been absent at baseline, or, if present at baseline, appears to have worsened in severity or frequency, regardless of its relation to the intervention. Adverse events deemed 'Possibly', 'Probably', or 'Definitely' related to the intervention were labeled as treatment-related adverse events (TRAE).
Time Frame: Up to 2 years
Population: Safety Population is defined as all participants who received at least 1 dose of any study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 6 | 8
Participants
  Treatment-related adverse event (TRAE) | 5 | 4
  Grade 3 or Grade 4 TRAE | 1 | 0
  Grade 5 TRAE | 0 | 0
  Serious TRAE | 1 | 0
  TRAE leading to treatment discontinuation | 1 | 0

2. Secondary Outcome: Mean Change From Baseline in the Number of Newly Appearing Spore-forming Species
Description: Engraftment was defined as the number of spore-forming species detected in SER-401 that were absent in participant baseline samples, and present post-microbiome-treatment, also referred to as newly appearing dose species.
Time Frame: Up to 2 years
Population: Participants were excluded from analysis at a specific time point if a stool sample was not collected or there was insufficient material available to run the assay.
Measure: Mean (Standard Deviation); unit: spore-forming species
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 6 | 8
spore-forming species
  Day -7: number analyzed (Participants) | 6 | 6
  Day -7 | 5.33 (7.202) | 1.67 (1.862)
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 7
  Cycle 1 Day 1 | 6.83 (8.424) | 25.71 (17.661)
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 7
  Cycle 1 Day 8 | 7.60 (9.209) | 23.29 (5.187)
  Cycle 2 Day 1 | 7.67 (10.539) | 28.38 (16.767)
  Cycle 3 Day 1: number analyzed (Participants) | 6 | 6
  Cycle 3 Day 1 | 8.50 (12.629) | 29.00 (12.853)
  Cycle 4 Day 1: number analyzed (Participants) | 5 | 4
  Cycle 4 Day 1 | 4.80 (1.483) | 21.25 (6.551)
  Cycle 7 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 7 Day 1 | 11.20 (18.349) | 25.33 (8.963)

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the proportion of participants who attain a best overall response of complete response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions), as determined by RECIST version 1.1. Confirmation of response by a repeat tumor assessment is not required.
Time Frame: Up to week 52
Measure: Count of Participants; unit: Participants
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 6 | 8
Participants | 4 | 2

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Defined as CR, PR, or stable disease (SD) for ≥ 24 weeks as best response by RECIST v1.1.
Time Frame: Up to week 52
Measure: Count of Participants; unit: Participants
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 6 | 8
Participants | 5 | 3

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from randomization to date of first documented progression of disease, date of death due to any cause, or date of most recent participant contact that documented progression-free status
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 6 | 8
month | 15 [3.3 to NA] — The upper limit of the 95% CI is not available due to an insufficient number of participants with an event. | 5.2 [2.2 to NA] — The upper limit of the 95% CI is not available due to an insufficient number of participants with an event.

6. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from randomization until death or last contact if still alive at the time of final data collection (after completion of anti-PD-1 therapy).
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 6 | 8
month | NA [13.7 to NA] — Median OS and the upper limit of the 95% CI are not available due to an insufficient number of participants with an event (i.e. death). | 21.1 [9.1 to NA] — The upper limit of the 95% CI is not available due to an insufficient number of participants with an event (i.e. death).

7. Secondary Outcome: Duration of Response
Description: Defined as time from date of documented CR or PR to date of first documented progression of disease, date of death due to any cause, or date of most recent participant contact that documented response (ie, scan date).
Time Frame: Up to 2 years
Population: The overall number of participants evaluated for duration of response includes only those who achieved a complete (CR) or partial response (PR) as per RECIST v1.1.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 4 | 2
month | NA [5.7 to NA] — Median duration of response and the upper limit of the 95% CI are not available due to an insufficient number of participants with an event. | NA [NA to NA] — Median duration of response and the upper and lower limits of the 95% CI are not available due to an insufficient number of participants with an event.

8. Secondary Outcome: Absolute Change in the Percentage of CD8 Cells in Tumor Tissue From Baseline at Cycle 2.
Description: Absolute change in the percentage of CD8 cells in tumor tissue from baseline at Cycle 2.
Time Frame: At cycle 2 (each cycle is 28 days)
Population: Only participants with available CD8 values at both baseline at Cycle 2 are included in the analysis.
Measure: Median (Full Range); unit: percentage of CD8 cells
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
Number analyzed (Participants) | 1 | 2
percentage of CD8 cells | 62.7 [62.7 to 62.7] | 27.1 [17.6 to 36.6]

ADVERSE EVENTS:
Time Frame: All AEs were collected from the start of the study intervention until 100 days after the last dose of the study intervention, up to 2 years. Deaths were collected up to 2 years from the initiation of study intervention.
Description: Serious Adverse Events and Other (Not Including Serious) Adverse Events include both treatment-related and non-treatment-related events.
Arm/Group | SER-401 Matching Placebo/ Nivolumab | SER-401/ Nivolumab
All-Cause Mortality (participants affected / at risk) | 1/6 | 4/8
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER-401 Matching Placebo/ Nivolumab (N=6) | SER-401/ Nivolumab (N=8)
Primary adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SER-401 Matching Placebo/ Nivolumab (N=6) | SER-401/ Nivolumab (N=8)
Fatigue (General disorders) | 5 | 6
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 1 | 0
Dental discomfort (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin weeping (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Phantom limb syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Rash pustular (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Tinea versicolour (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Nocturia (Renal and urinary disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Pallor (Vascular disorders) | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Mastoid disorder (Ear and labyrinth disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Wound drainage (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT03817125/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT03817125/SAP_001.pdf